CLINICAL TRIAL: NCT00848393
Title: Stress Response in Children Undergoing Cardiac Surgery: a Prospective Randomized Comparison Between Low Dose Fentanyl (LDF), Low Dose Fentanyl Plus Dexmedetomidine (LDF + Dex) and High Dose Fentanyl (HDF).
Brief Title: Measures to Lower the Stress Response in Pediatric Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Aymen N Naguib, Director of Pediatric Cardiothoracic Anesthesia, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB08-00029; 101911 (Other: FDA)
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Tetralogy of Fallot (TOF); Ventricular Septal Defects (VSD); Atrioventricular Septal Defects (AVSD)
Keywords: pediatric cardiac surgery; stress response; early extubation; Dexmedetomidine; TOF; VSD; AVSD
MeSH Terms: conditions — Tetralogy of Fallot; Heart Septal Defects, Ventricular; Endocardial Cushion Defects; Fractures, Stress; Atrioventricular Septal Defect | interventions — Fentanyl; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fentanyl (High Dose) (Active Comparator): This arm will receive a total of 25 mcg/kg of Fentanyl (High Dose) in two divided doses. First half-dose given at induction and second half-dose given before incision.
  Interventions: Drug: Fentanyl (High Dose)
- Fentanyl (Low Dose) (Active Comparator): This arm will receive a total of 10 mcg/kg of Fentanyl (Low Dose). First half-dose will be given at induction and second half -dose given before incision.
  Interventions: Drug: Fentanyl (Low Dose)
- Fentanyl (Low Dose) + Dexmedetomidine (Active Comparator): This arm will receive10 mcg/kg of Fentanyl (Low Dose) -2 divided doses. Dexmedetomidine (Dex) loading dose-1 mcg/kg over 10 min, then Dex infusion at 0.5mcg/kg/hr.
  Interventions: Drug: Fentanyl (Low Dose) + Dexmedetomidine

INTERVENTIONS:
Drug: Fentanyl (High Dose) — Fentanyl (High Dose) 25 mcg/kg in two divided doses. Half-dose will be given at induction and the second half-dose given prior to incision.
  Other Names: Fentanyl citrate
  Arms: Fentanyl (High Dose)
Drug: Fentanyl (Low Dose) — Fentanyl (Low Dose) 10 mcg/kg in two divided doses. Half-dose will be given at induction and the second half-dose given prior to incision.
  Other Names: Fentanyl citrate
  Arms: Fentanyl (Low Dose)
Drug: Fentanyl (Low Dose) + Dexmedetomidine — Fentanyl (Low Dose) + Dexmedetomidine. Dexmedetomidine at 1mcg/kg loading dose over 10 minutes, followed by an infusion at a rate of 0.5mcg/kg/hr. In addition, this group will receive a total of 10 mcg/kg Fentanyl (Low Dose). Half the dose will be given at induction and the second half before incision.
  Other Names: Fentanyl citrate + Precedex for dexmedetomidine
  Arms: Fentanyl (Low Dose) + Dexmedetomidine

SUMMARY:
Cardiac surgery induces a measurable stress response in patients which leads to increased morbidity and mortality post-operatively. Through clinical observation, anesthesiologists have determined that varying the combinations of anesthesia drugs used during surgery and just after reduces the stress response, and by extension, morbidity and mortality. However, only a few studies have explored this phenomenon scientifically.

DETAILED DESCRIPTION:
In this study, we aim to demonstrate comparatively that use of dexmedetomidine in addition to low dose narcotics reduces the stress response in cardiac surgical patients and results in less morbidity and mortality. Additionally, dexmedetomidine (Dex) should facilitate safe early extubation in pediatric cardiac patients, which results in decreased ventilator associated co-morbidities. Patients will be randomly assigned to three groups; one group will receive low dose fentanyl (LDF), one will receive low dose fentanyl with dexmedetomidine (LDF + Dex), and one will receive high dose fentanyl (HDF). Blood samples will be collected post-induction, post-sternotomy, after going on cardiopulmonary bypass, at the completion of surgery, and post-operatively to determine the patients' stress hormone levels. The patients will receive standard post-operative care, and clinical data collected as part of this care will be used to determine the incidence of morbidity and mortality. The results of the blood tests will be correlated with the incidence of morbidity and mortality to demonstrate the relative effectiveness of the different anesthesia methods.

Blood samples will be analyzed for the presence of the stress hormones cortisol, epinephrine, norepinephrine, adrenocorticotropic hormone (ACTH), Interleukin 8 (IL-8), TNF-alpha (Tumor Necrosis Factor), and nitrated albumin. Arterial blood gas, glucose and lactate levels, heart rate, blood pressure, use of vasoactive support, length of ventilator use, post-operative mortality, post-operative morbidity, length of Intensive Care Unit (ICU) stay, and length of hospital stay will be recorded.

Children previously enrolled in the surgery study will complete assessments of their cognitive ability, developmental status, and emotional and behavioral adjustment. For the neuro-developmental outcome follow up, Children's cognitive ability will be assessed using the Stanford-Binet Intelligence Scales, 5th Edition (SB5). The SB5 is a widely-used measure of intellectual functioning that is normed for ages 2 and up. The test takes 30-50 minutes to administer to young children, and provides an overall Intelligence Quotient (IQ) score, as well as scores for five primary factors of cognitive ability: Fluid Reasoning, Knowledge, Quantitative Reasoning, Visual-Spatial Processing; and Working Memory. The SB5 has demonstrated excellent reliability and validity.

ELIGIBILITY:
Inclusion Criteria:

* Childrens with the diagnosis of tetralogy of fallot, ventricular septal defect and atrioventricular septal defect who are under one year of age.

Exclusion Criteria:

* Patients who are having reoperation.
* Patients with comorbidities, such as heart failure.
* Patients receiving digoxin preoperatively.

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2008-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aymen N Naguib, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mukhtar AM, Obayah EM, Hassona AM. The use of dexmedetomidine in pediatric cardiac surgery. Anesth Analg. 2006 Jul;103(1):52-6, table of contents. doi: 10.1213/01.ane.0000217204.92904.76. PMID 16790625
- [Background] Mellon RD, Simone AF, Rappaport BA. Use of anesthetic agents in neonates and young children. Anesth Analg. 2007 Mar;104(3):509-20. doi: 10.1213/01.ane.0000255729.96438.b0. PMID 17312200
- [Background] Anand KJ, Hickey PR. Halothane-morphine compared with high-dose sufentanil for anesthesia and postoperative analgesia in neonatal cardiac surgery. N Engl J Med. 1992 Jan 2;326(1):1-9. doi: 10.1056/NEJM199201023260101. PMID 1530752
- [Background] Anand KJ, Hansen DD, Hickey PR. Hormonal-metabolic stress responses in neonates undergoing cardiac surgery. Anesthesiology. 1990 Oct;73(4):661-70. doi: 10.1097/00000542-199010000-00012. PMID 2221435
- [Background] Kapoor MC, Ramachandran TR. Inflammatory response to cardiac surgery and strategies to overcome it. Ann Card Anaesth. 2004 Jul;7(2):113-28. PMID 17827544
- [Background] Gruber EM, Laussen PC, Casta A, Zimmerman AA, Zurakowski D, Reid R, Odegard KC, Chakravorti S, Davis PJ, McGowan FX Jr, Hickey PR, Hansen DD. Stress response in infants undergoing cardiac surgery: a randomized study of fentanyl bolus, fentanyl infusion, and fentanyl-midazolam infusion. Anesth Analg. 2001 Apr;92(4):882-90. doi: 10.1097/00000539-200104000-00016. PMID 11273919

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 51 study subjects completed the study.
Pre-assignment Details: Total number of subjects recruited was 52 patients (one enrollee withdrew prior to any study-related procedures) resulting in a total number of subjects participating of 51. The enrollee was withdrawn from the study after signing the consent and prior to enrolling to one of the arms of the study.
Groups:
- Fentanyl (High Dose): Patients in this arm will receive a total of 25 mcg/kg of Fentanyl (High Dose) in two divided doses. first half will be given at induction and the second half will be given before incision.
  Fentanyl (High Dose): 25 mcg/kg in two divided doses. half the dose will be given at induction and the second half will be given prior to incision.
- Fentanyl (Low Dose): Patients in this arm will receive a total of 10 mcg/kg of Fentanyl (Low Dose). half the dose will be given at induction and the second half will be given before incision
  Fentanyl (Low Dose): patients will receive a total of 10 mcg/kg of Fentanyl (Low Dose). half the dose will be given at induction and the second half before incision.
- Fentanyl (Low Dose) + Dexmedetomidine: Patients in this arm will receive a total of 10 mcg/kg of Fentanyl (Low Dose) in two divided doses and Dexmedetomidine at a loading dose of 1 mcg/kg over 10 minutes and then an infusion of Dexmedetomidine at 0.5mcg/kg/hr.
  Fentanyl (Low Dose) + Dexmedetomidine: Dexmedetomidine at 1 mcg/kg loading dose over 10 minutes, followed by an infusion at a rate of 0.5 mcg/kg/hr. In addition, this group will receive a total of 10 mcg/kg Fentanyl (Low Dose). Half the dose will be given at induction and the second half before incision.
Period: Overall Study
Arm/Group | Fentanyl (High Dose) | Fentanyl (Low Dose) | Fentanyl (Low Dose) + Dexmedetomidine
Started | 17 | 16 | 18
Completed | 17 | 16 | 15
Not Completed | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — surgical complications unrelated to stud | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Fentanyl (Low Dose): patients in this group will receive a total of 10mcg/kg of fentanyl. half the dose will be given at induction and the second half will be given before incision
  Fentanyl (Low Dose): patients will receive a total of 10mcg/kg of fentanyl. half the dose will be given at induction and the second half before incision.
- Fentanyl (Low Dose) + Dexmedetomidine: patients in this group will receive a total of 10mcg/kg of Fentanyl (Low Dose) in two divided doses and Dexmedetomidine at a loading dose of 1mcg/kg over 10 minutes and then an infusion of Dexmedetomidine at 0.5mcg/kg/hr.
  Fentanyl (Low Dose) + Dexmedetomidine: Dexmedetomidine at 1mcg/kg loading dose over 10 minutes, followed by an infusion at a rate of 0.5mcg/kg/hr. In addition, this group will receive a total of 10 mcg/kg Fentanyl (Low Dose). Half the dose will be given at induction and the second half before incision.
- Total: Total of all reporting groups
Arm/Group | Fentanyl (High Dose) | Fentanyl (Low Dose) | Fentanyl (Low Dose) + Dexmedetomidine | Total
Number analyzed (Participants) | 17 | 16 | 15 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 16 | 15 | 48
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: months] | 4 [1 to 35] | 4 [3 to 7] | 5 [2 to 21] | 4 [1 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 4 | 16
  Male | 9 | 12 | 11 | 32
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 15 | 48

OUTCOME MEASURES:

1. Primary Outcome: ACTH and Cytokine Levels
Description: N = 48 n = 16 (LDF); n = 17 (HDF); n = 15 (LDF + Dex) ACTH assayed by enzyme-linked immunosorbent assay (ELISA); Cytokine levels in plasma were measured using the Immulite automated chemiluminometer. Measured cytokines include interleukin (IL)-6, IL-8, IL-10, and tumor necrosis factor-α.
Time Frame: Blood draws to measure cytokines levels within one hour of draw: after induction; after sternotomy; after starting cardiopulmonary bypass; at the end of the procedure; and 24 hours after the procedure.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Fentanyl (Low Dose): patients in this group will receive a total of 10mcg/kg of Fentanyl (Low Dose). half the dose will be given at induction and the second half will be given before incision
  Fentanyl (Low Dose): patients will receive a total of 10mcg/kg of Fentanyl (Low Dose). half the dose will be given at induction and the second half before incision.
- Fentanyl (Low Dose) + Dexmedetomidine: patients in this group will receive a total of 10mcg/kg of Fentanyl (Low Dose) in two divided doses and Dexmedetomidine at a loading dose of 1mcg/kg over 10 minutes and then an infusion of Dexmedetomidine at 0.5mcg/kg/hr.
  Fentanyl (Low Dose) + Dexmedetomidine: Dexmedetomidine at 1mcg/kg loading dose over 10 minutes, followed by an infusion at a rate of 0.5mcg/kg/hr.in addition this group will receive a total of 10 mcg/kg Fentanyl (Low Dose). Half the dose will be given at induction and the second half before incision.
Arm/Group | Fentanyl (High Dose) | Fentanyl (Low Dose) | Fentanyl (Low Dose) + Dexmedetomidine
Number analyzed (Participants) | 17 | 16 | 15
pg/mL
  Baseline ACTH (pg/mL) | 116.9 (117.0) | 182.7 (111.3) | 135.3 (129.8)
  Post-Sternotomy ACTH (pg/mL) | 44.5 (39.7) | 86.2 (76.5) | 106.9 (153.5)
  Post-Bypass ACTH (pg/mL) | 57.2 (61.2) | 172.7 (121.8) | 191.6 (220.2)
  End-Of-Surgery ACTH (pg/mL) | 66.4 (77.9) | 155.0 (107.5) | 154.1 (166.6)
  24 hour Post-Surgery ACTH (pg/mL) | 12.7 (7.4) | 53.2 (24.3) | 22.4 (130.3)
  Baseline TNF-alpha (pg/mL) | 15.70077 (16.401) | 25.294 (31.22396) | 8.018182 (10.68364)
  Post-Sternotomy TNF-alpha (pg/mL) | 26.51846 (33.64902) | 24.497 (33.8474) | 17.88636 (16.96651)
  Post-Bypass TNF-alpha (pg/mL) | 24.30615 (23.03753) | 25.787 (29.267) | 20.34364 (14.03041)
  End-Of-Surgery TNF-alpha (pg/mL) | 23.87077 (17.18903) | 24.857 (18.82328) | 23.06091 (18.8737)
  24 hour Post-Surgery TNF-alpha (pg/mL) | 15.79 (30.8563) | 11.954 (17.23623) | 21.13909 (19.00043)
  Baseline IL-6 (pg/mL) | 6.637058824 (4.356124661) | 4.757142857 (2.178819118) | 5.542857143 (3.455366904)
  Post-Sternotomy IL-6 (pg/mL) | 5.402353 (3.623996) | 12.17333 (28.79942) | 6.241333 (4.0798)
  Post-Bypass IL-6 (pg/mL) | 5.098824 (3.10355) | 5.509375 (3.93354) | 5.040667 (2.583747)
  End-Of-Surgery IL-6 (pg/mL) | 20.48571 (11.00962) | 22.47333 (12.59657) | 20.79231 (12.55537)
  24 hour Post-Surgery IL-6 (pg/mL) | 126.0813 (141.7456) | 117.975 (95.86805) | 142.1571 (129.4279)
  Baseline IL-8 (pg/mL) | 17.12353 (24.88048) | 10.44286 (1.839195) | 10.25714 (1.336306)
  Post-Sternotomy IL-8 (pg/mL) | 20.77647 (42.23163) | 10.66667 (2.941736) | 10.86667 (1.980861)
  Post-Bypass IL-8 (pg/mL) | 9.770588 (2.389499) | 10.13125 (2.15769) | 9.673333 (1.182894)
  End-Of-Surgery IL-8 (pg/mL) | 28.1 (17.28596) | 33.12667 (25.1446) | 37.22143 (43.66227)
  24 hour Post-Surgery IL-8 (pg/mL) | 49.07143 (69.39429) | 47.25 (99.4908) | 24.27143 (14.72541)
  Baseline IL-10 (pg/mL) | 10.82353 (1.952412) | 9.9 (0.00000) | 12.76429 (9.373252)
  Post-Sternotomy IL-10 (pg/mL) | 9.911765 (2.749291) | 9.9 (0.00000) | 14.10667 (13.63863)
  Post-Bypass IL-10 (pg/mL) | 9.488235 (1.872793) | 9.9 (2.581989) | 12.30667 (10.78136)
  End-Of-Surgery IL-10 (pg/mL) | 345.4412 (445.7443) | 325.55 (262.3603) | 569.2714 (858.2538)
  24 hour Post-Surgery IL-10 (pg/mL) | 10.80667 (1.907304) | 14.80833 (10.65888) | 9.692857 (0.775058)

2. Primary Outcome: Comparisons Between Groups for Narcotic and/or Dexmedetomidine Intervention Influence on Length of CTICU Stay.
Time Frame: Hospital admission to discharge from CTICU (average of 2-4 days)
Measure: Median (Full Range); unit: Days
Arm/Group | Fentanyl (High Dose) | Fentanyl (Low Dose) | Fentanyl (Low Dose) + Dexmedetomidine
Number analyzed (Participants) | 17 | 16 | 15
Days | 1 [1 to 8] | 1 [1 to 4] | 2 [1 to 5]

3. Primary Outcome: Comparisons Between Groups for Narcotic and/or Dexmedetomidine Intervention Influence on Time on Ventilator.
Time Frame: Time of intubation to extubation (variable)
Measure: Median (Full Range); unit: Hours
Arm/Group | Fentanyl (High Dose) | Fentanyl (Low Dose) | Fentanyl (Low Dose) + Dexmedetomidine
Number analyzed (Participants) | 17 | 16 | 15
Hours | 10.75 [0 to 27.32] | 3.79 [0 to 16] | 2.4 [0 to 2.4]

4. Primary Outcome: Stanford-Binet Intelligence Scales
Description: The Stanford-Binet test evaluates the overall IQ score from the assessment of cognitive ability. The test consists of 15 subtests, grouped into the four area scores. Six subtests are administered to all age levels. The subtests are: Vocabulary, Comprehension, Pattern Analysis, Quantitative, Bead Memory, and Memory for Sentences. Number of tests administered and test difficulty are based on the test taker's age and performance on subtest measuring word knowledge. The word knowledge subtest is given to all test takers and is the first subtest administered. A score of 100 is in the normal or average range. Higher scores suggest a higher level of functioning related to each category. (University of Cincinnati, 2003) Raw scores for each subtest within the overall test are converted to scaled scores using a table within each test manual to look up equivalents. Scaled scores are then converted to standard scores (range=50-150).
Time Frame: 1-4 yrs. post-surgery
Population: Six patients underwent their surgical repair after 1 y of age and were excluded from the follow-up neurodevelopmental testing post-surgery. 2 patients were deceased, 11 families refused to participate, 8 patients could not be reached due to relocation to other states or outside the country leaving a total of 21 patients.
Measure: Mean (Standard Deviation); unit: IQ
Arm/Group | Fentanyl (High Dose) | Fentanyl (Low Dose) | Fentanyl (Low Dose) + Dexmedetomidine
Number analyzed (Participants) | 5 | 9 | 7
IQ
  Nonverbal IQ composite score | 92 (19) | 98 (15) | 89 (6)
  Verbal IQ composite score | 93 (26) | 91 (17) | 80 (8)
  Full-scale IQ composite score | 93 (24) | 94 (15) | 83 (5)

5. Primary Outcome: Stress Hormone Levels
Description: Cortisol, epinephrine, and norepinephrine assayed by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Blood draws to measure stress hormone levels within one hour of draw: after induction; after sternotomy; after starting cardiopulmonary bypass; at the end of the procedure; and 24 hours after the procedure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Fentanyl (High Dose) | Fentanyl (Low Dose) | Fentanyl (Low Dose) + Dexmedetomidine
Number analyzed (Participants) | 17 | 16 | 15
ng/mL
  Baseline Norepinephrine | 13.32618 (10.1541) | 19.34153 (9.880667) | 19.45968 (13.08422)
  Post-Sternotomy Norepinephrine | 16.2606 (9.929948) | 17.08766 (8.419782) | 12.74458 (11.4669)
  Post-Bypass Norepinephrine | 23.35796 (13.54953) | 22.31064 (17.06955) | 19.73612 (17.07041)
  End-of-Surgery Norepinephrine | 11.22376 (8.599634) | 10.74731 (8.144776) | 7.727055 (13.04373)
  24 hour Post-Surgery Norepinephrine | 19.03031 (17.41692) | 20.85433 (18.38192) | 26.67379 (26.06332)
  Baseline ephinephrine | 2.7848 (3.127335) | 6.439221 (7.528216) | 5.876335 (9.551871)
  Post-Sternotomy Epinephrine | 2.376012 (2.273879) | 9.843591 (8.670264) | 10.89824 (16.85818)
  Post-Bypass Epinephrine | 18.176 (22.04968) | 21.9075 (15.02187) | 20.5294 (17.2838)
  End-of-Surgery Epinephrine | 14.65742 (18.34983) | 8.620669 (6.799042) | 8.083004 (8.808354)
  24 hour Post-Surgery Epinephrine | 5.004787 (6.666509) | 3.537063 (2.466451) | 4.418208 (6.764226)
  Baseline Cortisol | 334.7762 (314.6592) | 449.1974 (279.4671) | 352.4913 (265.2216)
  Post-Sternotomy Cortisol | 353.5396 (281.4853) | 363.5948 (164.9006) | 361.0074 (223.3172)
  Post-Bypass Cortisol | 279.0063 (188.1155) | 395.1298 (173.3926) | 354.8089 (210.7565)
  End-of-Surgery Cortisol | 333.0644 (294.8148) | 463.3857 (251.6977) | 387.3673 (191.7376)
  24 hour Post-Surgery Cortisol | 237.5506 (243.8181) | 266.8754 (239.2913) | 265.7373 (291.3256)

6. Secondary Outcome: Stanford-Binet Cognitive Ability
Description: The Stanford-Binet Intelligence Scale is now in its fifth edition (SB5) and was released in 2003. It is a cognitive ability and intelligence test that is used to diagnose developmental or intellectual deficiencies in young children. The test measures five weighted factors and consists of both verbal and nonverbal subtests. The five factors being tested are knowledge, quantitative reasoning, visual-spatial processing, working memory, and fluid reasoning. Raw scores for each subtest within the overall test are converted to scaled scores using a table within each test manual to look up equivalents. Scaled scores are then converted to standard scores (range=50-150). Higher scores suggest a higher level of functioning related to each category.
Time Frame: 1-4 yrs post-surgery
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fentanyl (High Dose) | Fentanyl (Low Dose) | Fentanyl (Low Dose) + Dexmedetomidine
Number analyzed (Participants) | 5 | 9 | 7
units on a scale
  Quantative Reasoning Score | 106 (22) | 96 (18) | 82 (15)
  Knowledge Score | 91 (27) | 97 (10) | 95 (12)
  Visual Spatial Processing Score | 91 (17) | 97 (16) | 92 (7)
  Working Memory Score | 94 (17) | 92 (10) | 84 (13)
  Fluid Reasoning Score | 86 (20) | 93 (19) | 75 (10)

7. Secondary Outcome: ABAS-II
Description: The ABAS-II is designed to evaluate whether an individual displays various functional skills necessary for daily living without the assistance of others. Thus, this instrument focuses on independent behaviors and measures what an individual actually does, in addition to measuring what he or she may be able to do. In addition, the ABAS-II focuses on behaviors an individual displays on his or her own, without assistance from others. The Parent/Primary Caregiver Form is a comprehensive, diagnostic measure of the adaptive skills that have primary relevance for the functioning of infants, toddlers, and preschoolers in the home and other settings, and can be completed by parents or other primary care providers. Each composite or domain score is determined by summing the appropriate scaled scores and then determining its equivalent composite or domain score by looking it up in a table located in the manual.The range for all scores is 50-150, with a higher score equaling a better outcome.
Time Frame: 1-4 yrs post-surgery
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fentanyl (High Dose) | Fentanyl (Low Dose) | Fentanyl (Low Dose) + Dexmedetomidine
Number analyzed (Participants) | 5 | 9 | 7
units on a scale
  ABAS-II General Adaptive Composite Score | 96 (21) | 102 (13) | 100 (13)
  ABAS-II Conceptual Adaptive Domain Score | 99 (21) | 106 (16) | 99 (13)
  ABAS-II Social Adaptive Domain Score | 102 (24) | 106 (8) | 105 (13)
  ABAS-II Practical Adaptive Domain Score | 93 (15) | 96 (14) | 95 (11)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each patient from start of surgical procedure until hospital discharge (Length of Hospital Stay averaging 5 Days).
Groups:
- Fentanyl (Low Dose) + Dexmedetomidine: patients in this group will receive a total of 10mcg/kg of fentanyl in two divided doses and Dexmedetomidine at a loading dose of 1mcg/kg over 10 minutes and then an infusion of Dexmedetomidine at 0.5mcg/kg/hr.
  Fentanyl (Low Dose) + Dexmedetomidine: Dexmedetomidine at 1mcg/kg loading dose over 10 minutes, followed by an infusion at a rate of 0.5mcg/kg/hr.in addition this group will receive a total of 10 mcg/kg Fentanyl (Low Dose). Half the dose will be given at induction and the second half before incision.
Arm/Group | Fentanyl (High Dose) | Fentanyl (Low Dose) | Fentanyl (Low Dose) + Dexmedetomidine
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 2/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 1/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fentanyl (High Dose) (N=17) | Fentanyl (Low Dose) (N=16) | Fentanyl (Low Dose) + Dexmedetomidine (N=18)
Morbidity (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fentanyl (High Dose) (N=17) | Fentanyl (Low Dose) (N=16) | Fentanyl (Low Dose) + Dexmedetomidine (N=18)
Unblinded (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size related to: study components conceived after completion of initial stress response study, declined participation, and loss to follow-up. Inability to obtain pre-surgical baseline neurodevelopmental evaluations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes